CLINICAL TRIAL: NCT03235050
Title: A Phase IIb, Randomised, Parallel, Double-Blind Placebo-Controlled and Open-Label Active Comparator Study to Evaluate the Efficacy and Safety of MEDI0382 in the Treatment of Overweight and Obese Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Efficacy and Safety of MEDI0382 in the Treatment of Overweight and Obese Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5670C00004
Record Dates: First submitted 2017-07-21; First posted 2017-08-01 (Actual); Results first posted 2020-07-20 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — cotadutide; Liraglutide

STUDY DESIGN:
Intervention Model Description: Randomised, parallel, double-blind, placebo-controlled study with an open-label active comparator.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study will be conducted in a double-blind fashion for MEDI0382 and placebo. The sponsor staff, the subjects, and the Investigators involved in the treatment of subjects or in the clinical evaluation of subjects will not be aware of the treatment received. Liraglutide will be provided in an open-label active comparator arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- MEDI0382 low dose + Metformin (Experimental): Drug: MEDI0382 low dose Drug: Metformin tablets, total daily dose of ≥1500 mg (unless only tolerated at a lower dose)
  Interventions: Drug: MEDI0382 low dose
- MEDI0382 mid dose + Metformin (Experimental): Drug: MEDI0382 mid dose Drug: Metformin tablets, total daily dose of ≥1500 mg (unless only tolerated at a lower dose)
  Interventions: Drug: MEDI0382 mid dose
- MEDI0382 high dose + Metformin (Experimental): Drug: MEDI0382 high dose Drug: Metformin tablets, total daily dose of ≥1500 mg (unless only tolerated at a lower dose)
  Interventions: Drug: MEDI0382 high dose
- Placebo + Metformin (Placebo Comparator): Drug: Placebo Drug: Metformin tablets, total daily dose of ≥1500 mg (unless only tolerated at a lower dose)
  Interventions: Drug: Placebo
- Liraglutide + Metformin (Active Comparator): Drug: Liraglutide Drug: Metformin tablets, total daily dose of ≥1500 mg (unless only tolerated at a lower dose)
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: MEDI0382 low dose — Pharmaceutical form: solution Route of administration: subcutaneous
  Arms: MEDI0382 low dose + Metformin
Drug: MEDI0382 mid dose — Pharmaceutical form: solution Route of administration: subcutaneous
  Arms: MEDI0382 mid dose + Metformin
Drug: MEDI0382 high dose — Pharmaceutical form: solution Route of administration: subcutaneous
  Arms: MEDI0382 high dose + Metformin
Drug: Placebo — Pharmaceutical form: solution Route of administration: subcutaneous
  Arms: Placebo + Metformin
Drug: Liraglutide — Pharmaceutical form: solution Route of administration: subcutaneous
  Arms: Liraglutide + Metformin

SUMMARY:
This study is designed to evaluate the dose range for MEDI0382 with respect to blood glucose control and weight loss effects, as well as to further explore the safety profile of MEDI0382

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Male and female subjects aged ≥ 18 years at screening
* Body mass index ≥ 25 kg/m2 at screening
* HbA1c range of 7.0% to 10.5% (inclusive) at screening
* Diagnosed with type-2 diabetes mellitus (T2DM) and treated with metformin (stable dose of ≥1500 mg/day or maximal tolerated dose) for at least 2 months prior to screening. Use of another glucose-lowering medication for up to 2 weeks in the 2 months prior to screening is acceptable
* Women of childbearing potential (WOCBP), not breastfeeding and using appropriate birth control to avoid pregnancy throughout the study and for up to 4 weeks after the last dose of investigational product (IP), with a negative pregnancy test within 72 hours prior to the start of IP

Exclusion Criteria:

* History of, or any existing condition that, in the opinion of the Investigator, would interfere with evaluation of the IP, put the subject at risk, influence the subject's ability to participate or affect the interpretation of the results of the study and/or any subject unable or unwilling to follow study procedures
* Any subject who has received another IP as part of a clinical study or a GLP-1 receptor agonist containing preparation within the last 30 days or 5 half lives of the drug (whichever is longer) at the time of screening
* Severe allergy/hypersensitivity to any of the proposed study treatments or excipients
* Symptoms of acutely decompensated blood glucose control, a history of type 1 diabetes mellitus or diabetic ketoacidosis, or if the subject has been treated with daily subcutaneous (SC) insulin for a period longer than 2 weeks within 90 days prior to screening
* Acute or chronic pancreatitis. Subjects with serum triglyceride concentrations above 1000 mg/dL (11 mmol/L) at screening
* Significant inflammatory bowel disease or other severe disease or surgery affecting the upper Gastrointestinal (GI) tract
* Significant hepatic disease
* Impaired renal function defined as estimated glomerular filtration rate (eGFR) ≤30 mL/minute/1.73m2 at screening
* Severely uncontrolled hypertension
* Unstable angina pectoris, myocardial infarction (MI), transient ischaemic attack (TIA), or stroke within 3 months prior to screening
* Severe congestive heart failure

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 834 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (98):
- United States (20):
  - Research Site, Birmingham, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Glendale, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Marietta, Georgia
  - Research Site, Evansville, Indiana
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Metairie, Louisiana
  - Research Site, Elkridge, Maryland
  - Research Site, Bridgeton, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Brooklyn, New York
  - Research Site, Morehead City, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greer, South Carolina
  - Research Site, Houston, Texas
  - Research Site, Plano, Texas
  - Research Site, Layton, Utah
  - Research Site, Arlington, Virginia
  - Research Site, Manassas, Virginia
- Bulgaria (10):
  - Research Site, Botevgrad
  - Research Site, Kozloduy
  - Research Site, Kyustendil
  - Research Site, Lukovit
  - Research Site, Petrich
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Stara Zagora
- Canada (13):
  - Research Site, Red Deer, Alberta
  - Research Site, Sherwood Park, Alberta
  - Research Site, Burlington, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Guelph, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Thornhill, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Lévis, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Saint-Marc-des-Carrieres, Quebec
- Czechia (8):
  - Research Site, Beroun
  - Research Site, Jílové u Prahy
  - Research Site, Pardubice
  - Research Site, Pilsen
  - Research Site, Plzen - Severni Predmesti
  - Research Site, Prague
  - Research Site, Praha Klanovice
  - Research Site, Uherské Hradiště
- Germany (16):
  - Research Site, Aschaffenburg
  - Research Site, Berlin
  - Research Site, Eschweiler
  - Research Site, Essen
  - Research Site, Gelnhausen
  - Research Site, Hamburg
  - Research Site, Hof
  - Research Site, Löhne
  - Research Site, Lübeck
  - Research Site, Magdeburg
  - Research Site, Mannheim
  - Research Site, Münster
  - Research Site, Oldenburg
  - Research Site, Pirna
  - Research Site, Rhaunen
  - Research Site, Villingen-Schwenningen
- Mexico (4):
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Veracruz
- Russia (10):
  - Research Site, Chelyabinsk
  - Research Site, Izhevsk
  - Research Site, Kemerovo
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Perm
  - Research Site, Saint Petersburg
  - Research Site, Vladikavkaz
  - Research Site, Volgograd
  - Research Site, Yekaterinburg
- Slovakia (17):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Dolný Kubín
  - Research Site, Levice
  - Research Site, Lučenec
  - Research Site, Malacky
  - Research Site, Námestovo
  - Research Site, Nitra
  - Research Site, Nové Mesto nad Váhom
  - Research Site, Prievidza
  - Research Site, Rimavská Sobota
  - Research Site, Rožňava
  - Research Site, Sabinov
  - Research Site, Trebišov
  - Research Site, Trenčín
  - Research Site, Trnava
  - Research Site, Žilina

REFERENCES:
- [Derived] Nahra R, Wang T, Gadde KM, Oscarsson J, Stumvoll M, Jermutus L, Hirshberg B, Ambery P. Effects of Cotadutide on Metabolic and Hepatic Parameters in Adults With Overweight or Obesity and Type 2 Diabetes: A 54-Week Randomized Phase 2b Study. Diabetes Care. 2021 Jun;44(6):1433-1442. doi: 10.2337/dc20-2151. Epub 2021 May 20. PMID 34016612
- See also: D5670C00004 SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5670C00004&attachmentIdentifier=d3772b2d-e5a9-4fef-b796-e371735f6b2d&fileName=D5670C00004_SAP_redacted.pdf&versionIdentifier=
- See also: D5670C00004 CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5670C00004&attachmentIdentifier=e91d84a4-416d-4262-aea8-98b99f6854c5&fileName=D5670C00004_CSP_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo / Metformin tablets, total daily dose of ≥1500 mg (unless only tolerated at a lower dose)
- Liraglutide: Liraglutide + Metformin tablets, total daily dose of ≥1500 mg (unless only tolerated at a lower dose)
- MEDI0382 100 mcg: MEDI0382(cotadutide) low dose / Metformin tablets, total daily dose of ≥1500 mg (unless only tolerated at a lower dose)
- MEDI0382 200 mcg: MEDI0382(cotadutide) mid dose / Metformin tablets, total daily dose of ≥1500 mg (unless only tolerated at a lower dose)
- MEDI0382 300 mcg: MEDI0382(cotadutide) high dose / Metformin tablets, total daily dose of ≥1500 mg (unless only tolerated at a lower dose)
Period: Overall Study
Arm/Group | Placebo | Liraglutide | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Started | 112 | 110 | 100 | 256 | 256
Completed | 108 | 105 | 96 | 242 | 245
Not Completed | 4 | 5 | 4 | 14 | 11
Not completed — Adverse Event | 0 | 0 | 1 | 4 | 1
Not completed — Death | 0 | 0 | 0 | 2 | 1
Not completed — Lost to Follow-up | 1 | 2 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 2 | 5 | 7
Not completed — Other reasons | 0 | 1 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- MEDI0382 100 mcg: MEDI0382 low dose / Metformin tablets, total daily dose of ≥1500 mg (unless only tolerated at a lower dose)
- MEDI0382 200 mcg: MEDI0382 mid dose / Metformin tablets, total daily dose of ≥1500 mg (unless only tolerated at a lower dose)
- MEDI0382 300 mcg: MEDI0382 high dose / Metformin tablets, total daily dose of ≥1500 mg (unless only tolerated at a lower dose)
- Total: Total of all reporting groups
Arm/Group | Placebo | Liraglutide | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg | Total
Number analyzed (Participants) | 112 | 110 | 100 | 256 | 256 | 834
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (9.5) | 55.5 (9.8) | 57.6 (9.9) | 57.3 (9.9) | 56.3 (10.2) | 56.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 60 | 57 | 147 | 129 | 448
  Male | 57 | 50 | 43 | 109 | 127 | 386
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 0 | 5 | 0 | 11
  Asian | 1 | 1 | 0 | 3 | 1 | 6
  Black or African American | 0 | 3 | 1 | 3 | 3 | 10
  White | 107 | 103 | 99 | 245 | 252 | 806
  Other | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: To assess the effect of 100, 200, 300 μg of cotadutide on HbA1c versus placebo
Time Frame: From baseline to 14 weeks
Population: ITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 112 | 100 | 256 | 256
percentage | -0.18 [-0.34 to -0.02] | -1.01 [-1.18 to -0.84] | -1.22 [-1.33 to -1.11] | -1.09 [-1.20 to -0.98]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382 100 mcg; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.83, 95% CI 2-sided [-1.06 to -0.59]
Statistical Analysis 2: Comparison: Placebo vs MEDI0382 200 mcg; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -1.04, 95% CI 2-sided [-1.23 to -0.85]
Statistical Analysis 3: Comparison: Placebo vs MEDI0382 300 mcg; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.91, 95% CI 2-sided [-1.11 to -0.72]

2. Primary Outcome: Percent Change in Body Weight
Description: To assess the effect of 100, 200, 300 μg of cotadutide on body weight versus placebo
Time Frame: From baseline to 14 weeks
Population: ITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 112 | 100 | 256 | 256
percentage | -0.70 [-1.44 to 0.04] | -2.70 [-3.49 to -1.91] | -3.47 [-3.95 to -2.98] | -4.33 [-4.82 to -3.84]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382 100 mcg; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.00, 95% CI 2-sided [-3.08 to -0.91]
Statistical Analysis 2: Comparison: Placebo vs MEDI0382 200 mcg; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.76, 95% CI 2-sided [-3.65 to -1.87]
Statistical Analysis 3: Comparison: Placebo vs MEDI0382 300 mcg; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -3.62, 95% CI 2-sided [-4.51 to -2.73]

3. Secondary Outcome: Change in HbA1c
Description: To assess the effect of 100, 200, 300 μg of cotadutide on HbA1c versus placebo
Time Frame: from baseline to 26 weeks and 54 weeks
Population: ITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 112 | 100 | 256 | 256
percentage
  from baseline to 26 weeks: number analyzed (Participants) | 112 | 98 | 252 | 252
  from baseline to 26 weeks | -0.40 [-0.58 to -0.22] | -1.06 [-1.25 to -0.87] | -1.22 [-1.34 to -1.10] | -1.12 [-1.24 to -1.00]
  from baseline to 54 weeks: number analyzed (Participants) | 112 | 98 | 252 | 252
  from baseline to 54 weeks | -0.44 [-0.63 to -0.24] | -0.96 [-1.16 to -0.75] | -1.06 [-1.19 to -0.93] | -1.01 [-1.14 to -0.88]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382 100 mcg; Week 26; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.66, 95% CI 2-sided [-0.92 to -0.40]
Statistical Analysis 2: Comparison: Placebo vs MEDI0382 200 mcg; Week 26; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.81, 95% CI 2-sided [-1.03 to -0.60]
Statistical Analysis 3: Comparison: Placebo vs MEDI0382 300 mcg; Week 26; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.72, 95% CI 2-sided [-0.94 to -0.51]
Statistical Analysis 4: Comparison: Placebo vs MEDI0382 100 mcg; Week 54; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-0.80 to -0.24]
Statistical Analysis 5: Comparison: Placebo vs MEDI0382 200 mcg; Week 54; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.63, 95% CI 2-sided [-0.86 to -0.39]
Statistical Analysis 6: Comparison: Placebo vs MEDI0382 300 mcg; Week 54; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -0.57, 95% CI 2-sided [-0.80 to -0.34]

4. Secondary Outcome: Percentage of Participants Achieving an HbA1c Target < 7.0%
Description: To assess the effect of 100, 200, and 300 μg of cotadutide on percentage of participants achieving an HbA1c target of <7% versus placebo
Time Frame: after 14, 26, and 54 weeks
Population: Intent-to-Treat (ITT) population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 112 | 100 | 256 | 256
Participants
  after 14 weeks: number analyzed (Participants) | 112 | 98 | 252 | 252
  after 14 weeks | 19 | 50 | 143 | 143
  after 26 weeks: number analyzed (Participants) | 112 | 98 | 252 | 252
  after 26 weeks | 25 | 48 | 139 | 143
  after 54 weeks: number analyzed (Participants) | 112 | 98 | 252 | 252
  after 54 weeks | 23 | 52 | 125 | 128
Statistical Analysis 1: Comparison: Placebo vs MEDI0382 100 mcg; Week 14; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 6.67, 92% CI 2-sided [3.34 to 13.30]
Statistical Analysis 2: Comparison: Placebo vs MEDI0382 200 mcg; Week 14; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 9.95, 95% CI 2-sided [5.39 to 18.36]
Statistical Analysis 3: Comparison: Placebo vs MEDI0382 300 mcg; Week 14; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 8.52, 95% CI 2-sided [4.65 to 15.61]
Statistical Analysis 4: Comparison: Placebo vs MEDI0382 100 mcg; Week 26; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 3.74, 95% CI 2-sided [1.98 to 7.03]
Statistical Analysis 5: Comparison: Placebo vs MEDI0382 200 mcg; Week 26; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 5.40, 95% CI 2-sided [3.13 to 9.34]
Statistical Analysis 6: Comparison: Placebo vs MEDI0382 300 mcg; Week 26; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 5.20, 95% CI 2-sided [3.02 to 8.97]
Statistical Analysis 7: Comparison: Placebo vs MEDI0382 100 mcg; Week 54; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 4.94, 95% CI 2-sided [2.61 to 9.36]
Statistical Analysis 8: Comparison: Placebo vs MEDI0382 200 mcg; Week 54; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 4.55, 95% CI 2-sided [2.62 to 7.89]
Statistical Analysis 9: Comparison: Placebo vs MEDI0382 300 mcg; Week 54; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 4.34, 95% CI 2-sided [2.51 to 7.51]

5. Secondary Outcome: Percent Change in Body Weight
Description: To assess the effect of 100, 200, and 300 μg of cotadutide on body weight versus placebo
Time Frame: from baseline to 26 weeks and 54 weeks
Population: ITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 112 | 100 | 256 | 256
percentage
  from baseline to 26 weeks: number analyzed (Participants) | 112 | 98 | 253 | 250
  from baseline to 26 weeks | -1.14 [-1.99 to -0.29] | -3.23 [-4.13 to -2.32] | -3.94 [-4.51 to -3.38] | -4.60 [-5.17 to -4.04]
  from baseline to 54 weeks: number analyzed (Participants) | 112 | 98 | 253 | 250
  from baseline to 54 weeks | -0.84 [-1.82 to 0.14] | -3.27 [-4.32 to -2.22] | -3.08 [-3.73 to -2.43] | -4.16 [-4.81 to -3.50]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382 100 mcg; Week 26; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.09, 95% CI 2-sided [-3.32 to -0.85]
Statistical Analysis 2: Comparison: Placebo vs MEDI0382 200 mcg; Week 26; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.80, 95% CI 2-sided [-3.82 to -1.79]
Statistical Analysis 3: Comparison: Placebo vs MEDI0382 300 mcg; Week 26; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -3.46, 95% CI 2-sided [-4.48 to -2.44]
Statistical Analysis 4: Comparison: Placebo vs MEDI0382 100 mcg; Week 54; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.43, 95% CI 2-sided [-3.86 to -1.00]
Statistical Analysis 5: Comparison: Placebo vs MEDI0382 200 mcg; Week 54; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.24, 95% CI 2-sided [-3.41 to -1.06]
Statistical Analysis 6: Comparison: Placebo vs MEDI0382 300 mcg; Week 54; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -3.32, 95% CI 2-sided [-4.49 to -2.14]

6. Secondary Outcome: Absolute Change in Body Weight
Description: To assess the effect of 100, 200, 300 μg of cotadutide on body weight versus placebo
Time Frame: from baseline to 14 weeks, 26 weeks and 54 weeks
Population: ITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 112 | 100 | 256 | 256
kg
  from baseline to 14 weeks: number analyzed (Participants) | 108 | 94 | 248 | 245
  from baseline to 14 weeks | -0.71 [-1.44 to 0.03] | -2.66 [-3.45 to -1.87] | -3.45 [-3.94 to -2.97] | -4.42 [-4.91 to -3.93]
  from baseline to 26 weeks: number analyzed (Participants) | 112 | 98 | 253 | 250
  from baseline to 26 weeks | -1.20 [-2.06 to -0.34] | -3.20 [-4.13 to -2.28] | -3.94 [-4.52 to -3.37] | -4.75 [-5.33 to -4.18]
  from baseline to 54 weeks: number analyzed (Participants) | 112 | 98 | 253 | 250
  from baseline to 54 weeks | -0.94 [-1.94 to 0.07] | -3.20 [-4.28 to -2.12] | -3.09 [-3.77 to -2.42] | -4.35 [-5.03 to -3.68]
Statistical Analysis 1: Comparison: Placebo vs MEDI0382 100 mcg; Week 14; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -1.95, 95% CI 2-sided [-3.03 to -0.87]
Statistical Analysis 2: Comparison: Placebo vs MEDI0382 200 mcg; Week 14; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.75, 95% CI 2-sided [-3.63 to -1.86]
Statistical Analysis 3: Comparison: Placebo vs MEDI0382 300 mcg; Week 14; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -3.71, 95% CI 2-sided [-4.60 to -2.82]
Statistical Analysis 4: Comparison: Placebo vs MEDI0382 100 mcg; Week 26; Test type: Superiority; p = 0.002, ANCOVA; LS Mean Difference = -2.01, 95% CI 2-sided [-3.27 to -0.74]
Statistical Analysis 5: Comparison: Placebo vs MEDI0382 200 mcg; Week 26; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.74, 95% CI 2-sided [-3.78 to -1.71]
Statistical Analysis 6: Comparison: Placebo vs MEDI0382 300 mcg; Week 26; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -3.55, 95% CI 2-sided [-4.59 to -2.52]
Statistical Analysis 7: Comparison: Placebo vs MEDI0382 100 mcg; Week 54; Test type: Superiority; p = 0.003, ANCOVA; LS Mean Difference = -2.27, 95% CI 2-sided [-3.74 to -0.79]
Statistical Analysis 8: Comparison: Placebo vs MEDI0382 200 mcg; Week 54; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.16, 95% CI 2-sided [-3.37 to -0.95]
Statistical Analysis 9: Comparison: Placebo vs MEDI0382 300 mcg; Week 54; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -3.42, 95% CI 2-sided [-4.63 to -2.20]

7. Secondary Outcome: Percent Change in Body Weight Versus Active Comparator
Description: To assess the effect of 100, 200, and 300 μg of cotadutide on body weight versus liraglutide 1.8 mg once daily
Time Frame: from baseline to 14 weeks, 26 weeks and 54 weeks
Population: ITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage
Groups:
- Liraglutide: Liraglutide / Metformin tablets, total daily dose of ≥1500 mg (unless only tolerated at a lower dose)
Arm/Group | Liraglutide | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 110 | 100 | 256 | 256
percentage
  Percent change at 14 weeks: number analyzed (Participants) | 106 | 94 | 248 | 245
  Percent change at 14 weeks | -3.40 [-4.14 to -2.65] | -2.70 [-3.49 to -1.91] | -3.47 [-3.95 to -2.98] | -4.33 [-4.82 to -3.84]
  Percent change at 26 weeks: number analyzed (Participants) | 110 | 98 | 253 | 250
  Percent change at 26 weeks | -4.12 [-4.98 to -3.27] | -3.23 [-4.13 to -2.32] | -3.94 [-4.51 to -3.38] | -4.60 [-5.17 to -4.04]
  Percent change at 54 weeks: number analyzed (Participants) | 110 | 98 | 253 | 250
  Percent change at 54 weeks | -3.20 [-4.19 to -2.21] | -3.27 [-4.32 to -2.22] | -3.08 [-3.73 to -2.43] | -4.16 [-4.81 to -3.50]
Statistical Analysis 1: Comparison: Liraglutide vs MEDI0382 100 mcg; Percent change at Week 14; Test type: Superiority; p = 0.211, ANCOVA; LS Mean Difference = 0.70, 95% CI 2-sided [-0.39 to 1.79]
Statistical Analysis 2: Comparison: Liraglutide vs MEDI0382 200 mcg; Percent change at Week 14; Test type: Superiority; p = 0.881, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.96 to 0.83]
Statistical Analysis 3: Comparison: Liraglutide vs MEDI0382 300 mcg; Percent change at Week 14; Test type: Superiority; p = 0.042, ANCOVA; LS Mean Difference = -0.93, 95% CI 2-sided [-1.82 to -0.04]
Statistical Analysis 4: Comparison: Liraglutide vs MEDI0382 100 mcg; Percent change at Week 26; Test type: Superiority; p = 0.158, ANCOVA; LS Mean Difference = 0.90, 95% CI 2-sided [-0.35 to 2.14]
Statistical Analysis 5: Comparison: Liraglutide vs MEDI0382 200 mcg; Percent change at Week 26; Test type: Superiority; p = 0.734, ANCOVA; LS Mean Difference = 0.18, 95% CI 2-sided [-0.85 to 1.20]
Statistical Analysis 6: Comparison: Liraglutide vs MEDI0382 300 mcg; Percent change at Week 26; Test type: Superiority; p = 0.357, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-1.51 to 0.54]
Statistical Analysis 7: Comparison: Liraglutide vs MEDI0382 100 mcg; Percent change at Week 54; Test type: Superiority; p = 0.921, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-1.51 to 1.37]
Statistical Analysis 8: Comparison: Liraglutide vs MEDI0382 200 mcg; Percent change at Week 54; Test type: Superiority; p = 0.847, ANCOVA; LS Mean Difference = 0.12, 95% CI 2-sided [-1.07 to 1.30]
Statistical Analysis 9: Comparison: Liraglutide vs MEDI0382 300 mcg; Percent change at Week 54; Test type: Superiority; p = 0.112, ANCOVA; LS Mean Difference = -0.96, 95% CI 2-sided [-2.15 to 0.22]

8. Secondary Outcome: Absolute Change in Body Weight Versus Active Comparator
Description: To assess the effect of 100, 200, and 300 μg of cotadutide on body weight versus liraglutide 1.8 mg once daily
Time Frame: from baseline to 14 weeks, 26 weeks and 54 weeks
Population: ITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Liraglutide | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 110 | 100 | 256 | 256
kg
  Absolute change at 14 weeks: number analyzed (Participants) | 106 | 94 | 248 | 245
  Absolute change at 14 weeks | -3.25 [-4.00 to -2.51] | -2.66 [-3.45 to -1.87] | -3.45 [-3.94 to -2.97] | -4.42 [-4.91 to -3.93]
  Absolute change at 26 weeks: number analyzed (Participants) | 110 | 98 | 253 | 250
  Absolute change at 26 weeks | -3.90 [-4.77 to -3.03] | -3.20 [-4.13 to -2.28] | -3.94 [-4.52 to -3.37] | -4.75 [-5.33 to -4.18]
  Absolute change at 54 weeks: number analyzed (Participants) | 110 | 98 | 253 | 250
  Absolute change at 54 weeks | -2.94 [-3.96 to -1.92] | -3.20 [-4.28 to -2.12] | -3.09 [-3.77 to -2.42] | -4.35 [-5.03 to -3.68]
Statistical Analysis 1: Comparison: Liraglutide vs MEDI0382 100 mcg; Absolute change at Week 14; Test type: Superiority; p = 0.284, ANCOVA; LS Mean Difference = 0.59, 95% CI 2-sided [-0.49 to 1.68]
Statistical Analysis 2: Comparison: Liraglutide vs MEDI0382 200 mcg; Absolute change at Week 14; Test type: Superiority; p = 0.658, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-1.09 to 0.69]
Statistical Analysis 3: Comparison: Liraglutide vs MEDI0382 300 mcg; Absolute change at Week 14; Test type: Superiority; p = 0.010, ANCOVA; LS Mean Difference = -1.17, 95% CI 2-sided [-2.06 to -0.27]
Statistical Analysis 4: Comparison: Liraglutide vs MEDI0382 100 mcg; Absolute change at Week 26; Test type: Superiority; p = 0.279, ANCOVA; LS Mean Difference = 0.70, 95% CI 2-sided [-0.57 to 1.97]
Statistical Analysis 5: Comparison: Liraglutide vs MEDI0382 200 mcg; Absolute change at Week 26; Test type: Superiority; p = 0.940, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-1.08 to 1.00]
Statistical Analysis 6: Comparison: Liraglutide vs MEDI0382 300 mcg; Absolute change at Week 26; Test type: Superiority; p = 0.110, ANCOVA; LS Mean Difference = -0.85, 95% CI 2-sided [-1.89 to 0.19]
Statistical Analysis 7: Comparison: Liraglutide vs MEDI0382 100 mcg; Absolute change at Week 54; Test type: Superiority; p = 0.730, ANCOVA; LS Mean Difference = -0.26, 95% CI 2-sided [-1.74 to 1.22]
Statistical Analysis 8: Comparison: Liraglutide vs MEDI0382 200 mcg; Absolute change at Week 54; Test type: Superiority; p = 0.804, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-1.38 to 1.07]
Statistical Analysis 9: Comparison: Liraglutide vs MEDI0382 300 mcg; Absolute change at Week 54; Test type: Superiority; p = 0.023, ANCOVA; LS Mean Difference = -1.41, 95% CI 2-sided [-2.63 to -0.19]

9. Secondary Outcome: Percentage of Participants Achieving Weight Loss of ≥5% and ≥10%
Description: To assess the effect of 100, 200, and 300 μg of cotadutide on percentage of subjects achieving weight loss of ≥5% and ≥10% versus placebo
Time Frame: after 14 weeks, 26 weeks and 54 weeks
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 112 | 100 | 256 | 256
Participants
  Participants with weight loss ≥5% at Wk 14 (LOCF): number analyzed (Participants) | 108 | 94 | 248 | 245
  Participants with weight loss ≥5% at Wk 14 (LOCF) | 3 | 18 | 65 | 92
  Participants with weight loss ≥5% at Wk 26 (LOCF): number analyzed (Participants) | 112 | 98 | 253 | 250
  Participants with weight loss ≥5% at Wk 26 (LOCF) | 11 | 28 | 76 | 110
  Participants with weight loss ≥5% at Wk 54 (LOCF): number analyzed (Participants) | 112 | 98 | 253 | 250
  Participants with weight loss ≥5% at Wk 54 (LOCF) | 14 | 34 | 71 | 98
  Participants with weight loss ≥10% at Wk 14 (LOCF): number analyzed (Participants) | 108 | 94 | 248 | 245
  Participants with weight loss ≥10% at Wk 14 (LOCF) | 0 | 6 | 15 | 20
  Participants with weight loss ≥10% at Wk 26 (LOCF): number analyzed (Participants) | 112 | 98 | 253 | 250
  Participants with weight loss ≥10% at Wk 26 (LOCF) | 1 | 7 | 28 | 27
  Participants with weight loss ≥10% at Wk 54 (LOCF): number analyzed (Participants) | 112 | 98 | 253 | 250
  Participants with weight loss ≥10% at Wk 54 (LOCF) | 2 | 11 | 21 | 32
Statistical Analysis 1: Comparison: Placebo vs MEDI0382 100 mcg; weight loss >=5% at Week 14; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 8.37, 95% CI 2-sided [2.38 to 29.43]
Statistical Analysis 2: Comparison: Placebo vs MEDI0382 200 mcg; weight loss >=5% at Week 14; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 12.46, 95% CI 2-sided [3.82 to 40.64]
Statistical Analysis 3: Comparison: Placebo vs MEDI0382 300 mcg; weight loss >=5% at Week 14; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 21.26, 95% CI 2-sided [6.55 to 68.97]
Statistical Analysis 4: Comparison: Placebo vs MEDI0382 100 mcg; weight loss >=5% at Week 26; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 3.68, 95% CI 2-sided [1.72 to 7.89]
Statistical Analysis 5: Comparison: Placebo vs MEDI0382 200 mcg; weight loss >=5% at Week 26; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 3.95, 95% CI 2-sided [2.00 to 7.78]
Statistical Analysis 6: Comparison: Placebo vs MEDI0382 300 mcg; weight loss >=5% at Week 26; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 7.28, 95% CI 2-sided [3.72 to 14.24]
Statistical Analysis 7: Comparison: Placebo vs MEDI0382 100 mcg; weight loss >=5% at Week 54; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 3.71, 95% CI 2-sided [1.84 to 7.45]
Statistical Analysis 8: Comparison: Placebo vs MEDI0382 200 mcg; weight loss >=5% at Week 54; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio, log = 2.73, 95% CI 2-sided [1.46 to 5.09]
Statistical Analysis 9: Comparison: Placebo vs MEDI0382 300 mcg; weight loss >=5% at Week 54; Test type: Superiority; p < 0.001, ANCOVA; Odds Ratio, log = 4.48, 95% CI 2-sided [2.42 to 8.30]
Statistical Analysis 10: Comparison: Placebo vs MEDI0382 100 mcg; weight loss >=10% at Week 26; Test type: Superiority; p = 0.048, Regression, Logistic; Odds Ratio, log = 8.47, 95% CI 2-sided [1.02 to 70.17]
Statistical Analysis 11: Comparison: Placebo vs MEDI0382 200 mcg; weight loss >=10% at Week 26; Test type: Superiority; p = 0.010, Regression, Logistic; Odds Ratio, log = 13.81, 95% CI 2-sided [1.85 to 102.91]
Statistical Analysis 12: Comparison: Placebo vs MEDI0382 300 mcg; weight loss >=10% at Week 26; Test type: Superiority; p = 0.012, Regression, Logistic; Odds Ratio, log = 13.09, 95% CI 2-sided [1.75 to 97.68]
Statistical Analysis 13: Comparison: Placebo vs MEDI0382 100 mcg; weight loss >=10% at Week 54; Test type: Superiority; p = 0.013, Regression, Logistic; Odds Ratio, log = 6.92, 95% CI 2-sided [1.49 to 32.07]
Statistical Analysis 14: Comparison: Placebo vs MEDI0382 200 mcg; weight loss >=10% at Week 54; Test type: Superiority; p = 0.032, Regression, Logistic; Odds Ratio, log = 4.98, 95% CI 2-sided [1.15 to 21.60]
Statistical Analysis 15: Comparison: Placebo vs MEDI0382 300 mcg; weight loss >=10% at Week 54; Test type: Superiority; p = 0.005, Regression, Logistic; Odds Ratio, log = 7.91, 95% CI 2-sided [1.86 to 33.64]

10. Secondary Outcome: Percentage of Participants Rescued or Discontinued for Lack of Glycaemic Control
Description: To assess the effect of 100, 200, and 300 μg of cotadutide on the requirement for additional blood glucose-lowering therapies versus placebo
Time Frame: at 14 weeks, 26 weeks and 54 weeks
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 112 | 100 | 256 | 256
Participants
  received rescue medication at 14 wks | 11 | 1 | 3 | 2
  received rescue medication at 26 wks | 20 | 3 | 8 | 6
  received rescue medication at 54 wks | 34 | 10 | 26 | 24
  discontinued study IP at 14 wks | 2 | 0 | 1 | 0
  discontinued study IP at 26 wks | 4 | 1 | 2 | 0
  discontinued study IP at 54 wks | 4 | 1 | 3 | 0
Statistical Analysis 1: Comparison: Placebo vs MEDI0382 100 mcg; received rescue medication at 14 wks; Test type: Superiority; p = 0.024, Regression, Logistic; Odds Ratio, log = 0.09, 95% CI 2-sided [0.01 to 0.73]
Statistical Analysis 2: Comparison: Placebo vs MEDI0382 200 mcg; received rescue medication at 14 wks; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 0.11, 95% CI 2-sided [0.03 to 0.40]
Statistical Analysis 3: Comparison: Placebo vs MEDI0382 300 mcg; received rescue medication at 14 wks; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 0.07, 95% CI 2-sided [0.02 to 0.33]
Statistical Analysis 4: Comparison: Placebo vs MEDI0382 100 mcg; received rescue medication at 26 wks; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio, log = 0.14, 95% CI 2-sided [0.04 to 0.48]
Statistical Analysis 5: Comparison: Placebo vs MEDI0382 200 mcg; received rescue medication at 26 wks; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 0.14, 95% CI 2-sided [0.06 to 0.34]
Statistical Analysis 6: Comparison: Placebo vs MEDI0382 300 mcg; received rescue medication at 26 wks; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 0.11, 95% CI 2-sided [0.04 to 0.28]
Statistical Analysis 7: Comparison: Placebo vs MEDI0382 100 mcg; received rescue medication at 54 wks; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 0.24, 95% CI 2-sided [0.11 to 0.53]
Statistical Analysis 8: Comparison: Placebo vs MEDI0382 200 mcg; received rescue medication at 54 wks; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 0.24, 95% CI 2-sided [0.13 to 0.44]
Statistical Analysis 9: Comparison: Placebo vs MEDI0382 300 mcg; received rescue medication at 54 wks; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio, log = 0.22, 95% CI 2-sided [0.12 to 0.41]
Statistical Analysis 10: Comparison: Placebo vs MEDI0382 200 mcg; discontinued IP at 14 wks; Test type: Superiority; p = 0.216, Regression, Logistic; Odds Ratio, log = 0.22, 95% CI 2-sided [0.02 to 2.43]
Statistical Analysis 11: Comparison: Placebo vs MEDI0382 100 mcg; discontinued IP at 26 wks; Test type: Superiority; p = 0.253, Regression, Logistic; Odds Ratio, log = 0.28, 95% CI 2-sided [0.03 to 2.52]
Statistical Analysis 12: Comparison: Placebo vs MEDI0382 200 mcg; discontinued IP at 26 wks; Test type: Superiority; p = 0.079, Regression, Logistic; Odds Ratio, log = 0.21, 95% CI 2-sided [0.04 to 1.19]
Statistical Analysis 13: Comparison: Placebo vs MEDI0382 100 mcg; discontinued IP at 54 wks; Test type: Superiority; p = 0.252, Regression, Logistic; Odds Ratio, log = 0.27, 95% CI 2-sided [0.03 to 2.50]
Statistical Analysis 14: Comparison: Placebo vs MEDI0382 200 mcg; discontinued IP at 54 wks; Test type: Superiority; p = 0.143, Regression, Logistic; Odds Ratio, log = 0.32, 95% CI 2-sided [0.07 to 1.47]

11. Secondary Outcome: Pharmacokinetic (PK) Endpoint: Trough Plasma Concentration (Cmin)
Description: To characterise the PK profile of 100, 200, and 300 μg of cotadutide
Time Frame: Time points at which outcome measure were assessed for plasma concentration were Weeks 1,2,6,10,14,18,22,26, and 54
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 0 | 100 | 256 | 256
ng/mL
  Week 1: number analyzed (Participants) | 0 | 67 | 179 | 170
  Week 1 |  | 2.68 (1.27) | 2.76 (1.88) | 2.77 (1.84)
  Week 2: number analyzed (Participants) | 0 | 69 | 180 | 168
  Week 2 |  | 2.66 (1.61) | 5.13 (3.23) | 5.18 (3.05)
  Week 6: number analyzed (Participants) | 0 | 69 | 192 | 177
  Week 6 |  | 2.75 (1.44) | 5.20 (3.57) | 7.77 (4.88)
  Week 10: number analyzed (Participants) | 0 | 71 | 181 | 172
  Week 10 |  | 3.18 (2.26) | 5.74 (4.23) | 8.23 (4.31)
  Week 14: number analyzed (Participants) | 0 | 72 | 184 | 178
  Week 14 |  | 3.79 (4.05) | 6.50 (5.26) | 9.71 (7.64)
  Week 18: number analyzed (Participants) | 0 | 69 | 180 | 169
  Week 18 |  | 4.58 (5.04) | 7.43 (6.43) | 10.8 (7.95)
  Week 22: number analyzed (Participants) | 0 | 70 | 177 | 168
  Week 22 |  | 4.63 (4.28) | 8.07 (7.01) | 11.5 (9.77)
  Week 26: number analyzed (Participants) | 0 | 69 | 183 | 167
  Week 26 |  | 4.39 (3.33) | 8.12 (7.31) | 12.9 (12.1)
  Week 54: number analyzed (Participants) | 0 | 69 | 180 | 166
  Week 54 |  | 4.58 (3.89) | 8.99 (9.22) | 13.2 (14.3)

12. Secondary Outcome: Immunogenicity Endpoint: Overall Antidrug Antibody (ADA) Incidence (Number and Percentage of Positive Partipants)
Description: To characterise the immunogenicity of 100, 200, and 300 μg of cotadutide
Time Frame: Baseline through 54-week treatment period and 28-day follow-up
Population: As-treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 112 | 100 | 256 | 256
Participants
  ADA positive at baseline: number analyzed (Participants) | 111 | 98 | 250 | 249
  ADA positive at baseline | 1 | 1 | 0 | 0
  ADA incidence: number analyzed (Participants) | 111 | 97 | 248 | 250
  ADA incidence | 3 | 55 | 152 | 155
  ADA positive post-baseline: number analyzed (Participants) | 111 | 97 | 248 | 250
  ADA positive post-baseline | 3 | 54 | 152 | 155

13. Secondary Outcome: Immunogenicity Endpoint: Median Titer of the Anti-Drug Antibodies (ADA) to MEDI0382 in the Positive Participants
Description: To characterise the immunogenicity of 100, 200, and 300 μg of cotadutide
Time Frame: Baseline through 54-week treatment period and 28-day follow-up
Population: As-treated population
Measure: Median (Full Range); unit: titer
Arm/Group | Placebo | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
Number analyzed (Participants) | 112 | 100 | 256 | 256
titer
  ADA positive at baseline, median titer: number analyzed (Participants) | 111 | 98 | 250 | 249
  ADA positive at baseline, median titer | 5.0 [5 to 5] | 5.0 [5 to 5] | 0 [0 to 0] | 0 [0 to 0]
  ADA incidence, median of maximum titer: number analyzed (Participants) | 111 | 97 | 248 | 250
  ADA incidence, median of maximum titer | 5.0 [5 to 20] | 20.0 [5 to 2560] | 20.0 [5 to 640] | 20.0 [5 to 5120]
  ADA positive post-baseline, median of max. titer: number analyzed (Participants) | 111 | 97 | 248 | 250
  ADA positive post-baseline, median of max. titer | 5.0 [5 to 20] | 20.0 [5 to 2560] | 20.0 [5 to 640] | 20.0 [5 to 5120]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of first IP dose throughout the 54-week treatment period and including the 28-day follow-up period. Serious AEs were recorded from the time of signature of informed consent.
Arm/Group | Placebo | Liraglutide | MEDI0382 100 mcg | MEDI0382 200 mcg | MEDI0382 300 mcg
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/110 | 0/100 | 2/256 | 1/256
Serious Adverse Events (participants affected / at risk) | 12/112 | 8/110 | 12/100 | 33/256 | 20/256
Other Adverse Events (participants affected / at risk) | 45/112 | 36/110 | 51/100 | 159/256 | 164/256
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=112) | Liraglutide (N=110) | MEDI0382 100 mcg (N=100) | MEDI0382 200 mcg (N=256) | MEDI0382 300 mcg (N=256)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Silent myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Megacolon (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Post procedural fistula (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Triple negative breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo cns origin (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perinephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acquired phimosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vocal cord dysfunction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=112) | Liraglutide (N=110) | MEDI0382 100 mcg (N=100) | MEDI0382 200 mcg (N=256) | MEDI0382 300 mcg (N=256)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (3) | 1 (1) | 10 (10) | 13 (14)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 4 (7) | 13 (15) | 49 (68) | 28 (40)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 3 (3) | 7 (13) | 19 (26) | 28 (38)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 14 (17) | 12 (15)
Nausea (Gastrointestinal disorders) | 12 (13) | 17 (21) | 23 (28) | 85 (115) | 105 (143)
Vomiting (Gastrointestinal disorders) | 5 (6) | 3 (3) | 10 (12) | 51 (66) | 43 (58)
Nasopharyngitis (Infections and infestations) | 15 (19) | 11 (13) | 11 (13) | 22 (28) | 28 (44)
Respiratory tract infection viral (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 13 (15) | 7 (8)
Urinary tract infection (Infections and infestations) | 6 (6) | 2 (2) | 3 (4) | 13 (17) | 7 (9)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3) | 12 (12) | 14 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) | 8 (8) | 9 (12) | 9 (9)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 4 (5) | 11 (12) | 15 (19)
Headache (Nervous system disorders) | 1 (1) | 5 (5) | 3 (4) | 15 (18) | 19 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator shall provide AstraZeneca with copies of any materials relating to the Study, the Study Documentation, or the Developed Technologies that either Party intends to publish (or submit for publication) or make any presentations relating to, at least 60 days in advance of publication, submission or presentation.

DOCUMENTS (2):
  • Study Protocol (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/50/NCT03235050/Prot_002.pdf
  • Statistical Analysis Plan (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT03235050/SAP_003.pdf